CLINICAL TRIAL: NCT07291453
Title: Loving Habits: A Feasibility Study of a Support Program for Building New Parent-child Behavioral Habits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Okinawa Institute of Science and Technology Graduate University (Other)
Responsible Party: Principal Investigator, Emi Furukawa, Senior Staff Scientist, Okinawa Institute of Science and Technology Graduate University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR-2025-003
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Following-through module (Experimental): Parents will receive information about strategies during situations requiring following through on/completing tasks
  Interventions: Behavioral: Behavioral Parent Training
- Waiting module (Experimental): Parents will receive information about strategies during situations requiring waiting
  Interventions: Behavioral: Behavioral Parent Training
- Overcoming challenges module (Experimental): Parents will receive information about strategies during situations where a child finds it challenging to engage in tasks/behaviors, due to the the difficulty level or past failure
  Interventions: Behavioral: Behavioral Parent Training
- Transition module 1 (Experimental): Parents will receive information about strategies during situations where a child transitions from a preferred activity to a non-preferred activity over six videos.
  Interventions: Behavioral: Behavioral Parent Training
- Transition module 2 (Experimental): Parents will receive information about strategies during situations where a child transitions from a preferred activity to a non-preferred activity over two videos.
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Teaches parents antecedent- and reinforcement-based behavior management techniques and provide support to manage their stress

SUMMARY:
This study evaluates the feasibility and preliminary impacts of a new parent support program consisting of a series of educational videos, automatically delivered via a popular texting platform. The program content is focused on teaching parents strategies to better manage interactions with children in challenging situations many children experience, e.g., a transition to a non-preferred activity, waiting for delayed reward. Parents with children demonstrating inattentive, hyperactive and impulsive behavior and experiencing difficulties with these daily challenges are invited to participate in the study.

DETAILED DESCRIPTION:
This study employs a pre-post, open trial design with the primary aim to investigate the feasibility of delivering parenting educational materials in an accessible format, i.e., a widely used messaging platform. The training videos demonstrate the applications of antecedent- and reinforcement-based behavior management techniques in a specific situation and encourage parents to build positive parenting habits. The program usability and satisfaction will be assessed through participant ratings. The study targets parents of children demonstrating inattention, hyperactive, and impulsive behavior. These families frequently experience difficulties managing everyday routines at home, yet the access to psychosocial treatment is limited. The investigators expect parents to engage well in the program delivered via digital media. Based on the existing literature on the effectiveness of behavior parent training delivered in traditional in-person format, a moderate effect size is expected in the pre-post measures of parenting practices and the child target behavior for this study.

ELIGIBILITY:
Inclusion Criteria:

- Parents with children aged 4-10 who experience difficulties in situations targeted by the program.

*Note: The program will be advertised that it was developed targeting children demonstrating behaviors consistent with ADHD, and the ADHD symptoms will be measured pre-post. However, children are not required to have a diagnosis of ADHD or show elevated levels of ADHD symptoms for the mothers to sign up.

Exclusion Criteria:

- Parents who do not understand Japanese (the language the program is offered in).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-10-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of videos viewed | 1 month
  The number of videos viewed (minimum 0, maximum 6) to evaluate participant engagement.
Percentage of completed daily ratings | 1 month
  The percentage of completed daily ratings (minimum 0, maximum 100). Parents are asked to provide daily ratings on the degree of success in implementing parenting strategies taught.
Participant satisfaction | 1 month
  The parent-rated satisfaction regarding information presented in the videos. A rating completed after each video viewing using a 4-point scale. Averaged across the ratings completed for the videos viewed. (Minimum 0, maximum 4). Higher scores indicate greater satisfaction.

SECONDARY OUTCOMES:
Parent-rated child's difficulties in target situations | 1 month
  The parent-rated child's difficulties with daily target situation examples. Ratings completed before and after the intervention using a 4-point scale. Averaged across the ratings completed for the 7-9 situations (varies depending on the module). Higher scores indicate greater difficulties.
Parent-rated child's impairment related to target situations | 1 month
  The parent-rated level of impairment caused by transition difficulties (1 item). Ratings completed before and after the intervention using a 10 point scale. Lower scores indicate greater impairment.
Positive parenting | 1 month
  Positive and Negative Parenting Scale (PNPS) Positive Parenting sub-scale. Parent ratings completed before and after the intervention using a 4-point scale. Average across 4 items. Higher scores indicate more frequent use of positive parenting strategies.
Negative parenting | 1 month
  Description: Positive and Negative Parenting Scale (PNPS) Negative Parenting sub-scale. Parent ratings completed before and after the intervention using a 4-point scale. Average across 4 items. Higher scores indicate more frequent use of negative parenting strategies.
Parenting stress | 1 month
  Parent Stress Scale total score. Parent ratings completed before and after the intervention using a 5-point scale. Average across 10 items. Higher scores indicate higher levels of parent stress.

OTHER OUTCOMES:
ADHD symptoms | 1 month
  SNAP-IV inattention and hyperactivity/impulsivity symptoms total. Parent ratings completed before and after the intervention using a 4-point scale. Averaged across 18 items. Higher scores indicate ADHD symptoms more frequently observed.
ODD symptoms | 1 month
  SNAP-IV oppositional/defiant symptoms total. Parent ratings completed before and after the intervention using a 4-point scale. Averaged across 8 items. Higher scores indicate ADHD symptoms more frequently observed.

CONTACTS AND LOCATIONS:
Locations (1):
- Okinawa Institute of Science and Technology Graduate University, Onna, Okinawa, Japan

IPD SHARING:
Plan to Share IPD: No